CLINICAL TRIAL: NCT01745341
Title: Rates of Apnea in Patients Undergoing Vitreoretinal Surgery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Theodore Leng, Clinical Assistant Professor of Ophthalmology, Stanford University
Other Study IDs: 25284
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- vitreoretinal surgery patients: Patients undergoing vitreoretinal surgery under monitored anesthesia care. They will be observed during surgery and no interventions will be administered.

SUMMARY:
The purpose of this study is to determine if apnea (the stopping of breathing) occurs in patients undergoing undergoing monitored anesthesia care (MAC) for vitreoretinal surgery

DETAILED DESCRIPTION:
Patients undergoing vitreoretinal surgery will be monitored during the procedure to determine if they stop breathing. This study is observational in nature and no interventions will be made.

ELIGIBILITY:
Inclusion Criteria:

* patients having vitreoretinal surgery under monitored anesthesia care

Exclusion Criteria:

* patients having vitreoretinal surgery without monitored anesthesia care

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having vitreoretinal surgery under monitored anesthesia care
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Apnea | 15 minutes
  Determine if patients undergoing vitreoretinal surgery under monitored anesthesia care stop breathing during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States